CLINICAL TRIAL: NCT00576576
Title: The Evaluation of Atorvastatin on Wall Shear Stress, Atherosclerosis Composition, and Microvascular Function in Patients With Moderate Coronary Disease
Brief Title: Evaluation of Atorvastatin on Atherosclerosis Composition
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Emory University (Other)
Collaborators: Pfizer (Industry)
Responsible Party: Principal Investigator, Habib Samady, MD, Emory University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB00000701; GA2580TT (Other: Other); Emory #07052168 (Other: Other)
Record Dates: First submitted 2007-12-17; First posted 2007-12-19 (Estimated); Results first posted 2013-10-18 (Estimated); Last update posted 2013-12-24 (Estimated); Status verified 2013-11

CONDITIONS: Atherosclerosis
Keywords: Atherosclerosis, vulnerable plaque, IVUS, shear stress
MeSH Terms: conditions — Atherosclerosis | interventions — Atorvastatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- A (Experimental): All patients in this arm are given atorvastatin therapy.
  Interventions: Drug: Atorvastatin

INTERVENTIONS:
Drug: Atorvastatin — Atorvastatin 80 mg a day

SUMMARY:
The purpose of this study is to evaluate the effects of Atorvastatin on the coronary atherosclerosis plaque morphology.

DETAILED DESCRIPTION:
The primary goal of this project is to evaluate the effect of the cholesterol lowering drug Atorvastatin on the composition and character of coronary atherosclerosis (heart blockages). Atorvastatin is known to reduce cholesterol, reduce cardiac events, and halt the progression of coronary atherosclerosis. However, the reduction in cardiac events is out of proportion to the reductions in the total amount of atherosclerosis. Thus, the drug likely decreases cardiac events by changing the composition of the coronary atherosclerotic plaques. It is likely that the drug causes the "heart blockage" to change from a "vulnerable plaque" to a "stable" plaque. There are several features of "vulnerable plaques" that can be detected in arteries of the heart using intravascular ultrasound. The goal of this project is to examine the effects of atorvastatin on atherosclerosis plaque composition using this intravascular ultrasound in patients undergoing serial cardiac catheterizations. Our hypothesis is that atorvastatin will reduce the number of "vulnerable plaques" and increase the number of "stable plaques" seen by intravascular ultrasound. We plan to enroll a total of 20 patients. The patients will be evaluated by cardiac catheterization with intravascular ultrasound analysis and then be treated with atorvastatin for 6 months. These 20 patients will return to the cardiac catheterization laboratory 6 months later for a repeat catheterization with intravascular ultrasound evaluation.

The secondary goal of this proposal is to evaluate in humans the relationship between coronary atherosclerosis (plaque buildup in the arteries of the heart) and wall shear stress (the force generated against the wall of the artery by the flow of blood). The reason for this sub-study is that there is great interest in understanding the characteristics that cause the progression of coronary atherosclerosis. Local forces such as shear stress may play an important role in the focal progression of "vulnerable" atherosclerotic plaques. Indeed, low shear stress is known to be an important factor in the early formation of atherosclerosis. However, the relationship of low shear stress to development and progression of advanced "rupture prone" ("vulnerable") plaques has not been elucidated. Our hypotheses are: (1) "Vulnerable plaques" are more commonly located at areas of low shear stress(2) "Vulnerable plaques" at areas of low shear stress are more likely to progress over the following 6 months than plaques located in normal shear stress regions.

ELIGIBILITY:
Inclusion Criteria:

1. The patients are eligible if they are undergoing catheterization for stable angina or acute coronary syndromes
2. At the time of catheterization the patient has a "moderate coronary" lesion in the proximal 60mm of an epicardial coronary artery
3. "Moderate lesion" is defined as a lesion deemed significant enough to warrant further evaluation using coronary flow reserve (CFR) and fractional flow reserve (FFR) by the treating physician
4. Patient must have decision making capacity and consented prior to the catheterization
5. Ages: All ages
6. Performance Status: all levels

Exclusion Criteria:

1. Screening Exclusion Criteria:

1. Patients with coronary bypass grafts
2. Severe valvular heart disease
3. Patients presenting with a ST segment elevation myocardial infarction (STEMI)
4. Inability to provide informed consent prior to randomization
5. Creatinine >1.5
6. Patients who are on a statin with an LDL < 130.
7. Any patient on a maximum dose of statin (atorvastatin 80mg, simvastatin 80mg, rosuvastatin 20mg, pravastatin 80mg, or fluvastatin 80mg)
8. Uncontrolled diabetes requiring intensification of therapy
9. Uncontrolled hypertension requiring the addition of angiotensin-converting enzyme inhibitor or angiotensin receptor blocker

2. Angiographic Ineligibility Criteria:

1. A Left Main lesion greater than 50% stenosis
2. The moderate lesion is located beyond 60mm
3. Collaterals
4. Coronary Anatomy requiring coronary artery bypass grafting (CABG)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2007-07; Primary Completion 2010-03 (Actual); Study Completion 2010-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Habib Samady, MD, Principal Investigator — Emory University
Locations (1):
- Emory University Hospital, Atlanta, Georgia, United States

REFERENCES:
- [Background] Kawasaki M, Sano K, Okubo M, Yokoyama H, Ito Y, Murata I, Tsuchiya K, Minatoguchi S, Zhou X, Fujita H, Fujiwara H. Volumetric quantitative analysis of tissue characteristics of coronary plaques after statin therapy using three-dimensional integrated backscatter intravascular ultrasound. J Am Coll Cardiol. 2005 Jun 21;45(12):1946-53. doi: 10.1016/j.jacc.2004.09.081. PMID 15963391
- [Result] Samady H, Eshtehardi P, McDaniel MC, Suo J, Dhawan SS, Maynard C, Timmins LH, Quyyumi AA, Giddens DP. Coronary artery wall shear stress is associated with progression and transformation of atherosclerotic plaque and arterial remodeling in patients with coronary artery disease. Circulation. 2011 Aug 16;124(7):779-88. doi: 10.1161/CIRCULATIONAHA.111.021824. Epub 2011 Jul 25. PMID 21788584
- [Result] Eshtehardi P, McDaniel MC, Suo J, Dhawan SS, Avati Nanjundappa RP, Sawaya FJ, King AR, Oshinski JN, Taylor WR, Quyyumi AA, Giddens DP, Samady H. Coronary Plaque Progression Occurs Distal to Stenoses in Segments with Low Wall Shear Stress: A Prospective Evaluation in Patients with Coronary Artery Disease. Arterioscler Thromb Vasc Biol 2010;30(11);e251.
- [Derived] Eshtehardi P, McDaniel MC, Dhawan SS, Binongo JN, Krishnan SK, Golub L, Corban MT, Raggi P, Quyyumi AA, Samady H. Effect of intensive atorvastatin therapy on coronary atherosclerosis progression, composition, arterial remodeling, and microvascular function. J Invasive Cardiol. 2012 Oct;24(10):522-9. PMID 23043036

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 27 subjects enrolled and followed up for 6 months All subjects were recruited between 2007 and 2009 at Emory University Hospital
Groups:
- Atorvastatin: All patients in this arm are given atorvastatin therapy.
  Atorvastatin : Atorvastatin 80 mg a day
Period: Overall Study
Arm/Group | Atorvastatin
Started | 27
Completed | 20
Not Completed | 7
Not completed — Lost to Follow-up | 6
Not completed — Protocol Violation | 1

BASELINE CHARACTERISTICS:
Arm/Group | Atorvastatin
Number analyzed (Participants) | 20
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 14
  >=65 years | 6
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 54 (46-68) [46 to 68]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7
  Male | 13
Region of Enrollment [Number; unit: participants]
  United States | 20

OUTCOME MEASURES:

1. Primary Outcome: Change in Necrotic Core Volume
Description: Virtual Histology-Intravascular Ultrasound (VH-IVUS) defined necrotic core cross sectional area (CSA) measured in each VH-IVUS frame and averaged over length of studied vessel at baseline and follow -up. Change in necrotic core CSA between baseline and follow-up was calculated (subtracting the baseline value from the follow-up value).
Time Frame: 6 months
Population: All enrolled patients with complete data set
Measure: Mean (Standard Deviation); unit: mm^2
Arm/Group | Atorvastatin
Number analyzed (Participants) | 20
mm^2 | 0.07 (0.06)

2. Secondary Outcome: Change in Atheroma Volume
Description: Change in atheroma volume between baseline and follow-up is reported. This was derived by subtracting the baseline value from the 6-month value.
Time Frame: 6 months
Population: All enrolled patients with complete data set
Measure: Median (Inter-Quartile Range); unit: mm^3
Arm/Group | Atorvastatin
Number analyzed (Participants) | 20
mm^3 | -4.0 [-20.4 to 11.6]

3. Secondary Outcome: Change in Fibrous Plaque Volume
Description: Change in fibrous plaque volume between baseline and follow-up. This was derived by subtracting the baseline value from the 6-month value.
Time Frame: 6 months
Population: All enrolled patients with complete data set
Measure: Median (Inter-Quartile Range); unit: mm^3
Arm/Group | Atorvastatin
Number analyzed (Participants) | 20
mm^3 | -3.3 [-15.2 to 8.3]

ADVERSE EVENTS:
Arm/Group | Atorvastatin
Serious Adverse Events (participants affected / at risk) | 0/27
Other Adverse Events (participants affected / at risk) | 0/27

LIMITATIONS AND CAVEATS:
No adverse events to report.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No